CLINICAL TRIAL: NCT02964559
Title: A Phase II Trial of Pembrolizumab (MK-3475) in Metastatic Cutaneous Squamous Cell Carcinoma
Brief Title: Pembrolizumab in Patients With Locally Advanced or Metastatic Skin Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Michael Lowe, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00087412; NCI-2016-00831 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); Winship3185-16 (Other: Emory University/Winship Cancer Institute); P30CA138292 (NIH)
Record Dates: First submitted 2016-11-07; First posted 2016-11-16 (Estimated); Results first posted 2024-06-26 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Recurrent Skin Carcinoma; Skin Squamous Cell Carcinoma
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (pembrolizumab) (Experimental): Patients receive pembrolizumab IV over 30 minutes on day 1. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Pembrolizumab

INTERVENTIONS:
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475

SUMMARY:
This phase II trial studies how well pembrolizumab works in treating patients with skin cancer that has spread from where it started to nearby tissue, lymph nodes, or other parts of the body. Monoclonal antibodies, such as pembrolizumab, may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

-To establish the response rate of pembrolizumab in metastatic cutaneous squamous cell carcinoma.

SECONDARY OBJECTIVES:

-To determine the 6-month progression-free survival and 1 year overall survival of metastatic cutaneous squamous cell carcinoma of the skin (cSCC) treated with pembrolizumab.

OUTLINE:

Patients receive pembrolizumab intravenously (IV) over 30 minutes on day 1. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then every 8-12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* All subjects must have cutaneous squamous cell carcinoma that is not curable by surgery or radiation; both locally advanced and metastatic squamous cell carcinoma will be included.
* Be willing and able to provide written informed consent/assent for the trial.
* Have measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
* Be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion. Newly-obtained is defined as a specimen obtained up to 6 weeks (42 days) prior to initiation of treatment on day 1. Subjects for whom newly-obtained samples cannot be provided (e.g. inaccessible or subject safety concern) may submit an archived specimen only upon agreement from the sponsor.
* Be willing to undergo normal skin biopsy prior to initiation of treatment and after treatment.
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) performance scale.
* Absolute neutrophil count (ANC) ≥ 1,500/microliter (mcL)
* Platelets ≥ 100,000/mcL
* Hemoglobin ≥ 9 g/dL or ≥ 5.6 mmol/L without transfusion or erythropoietin (EPO) dependency (within 7 days of assessment)
* Serum creatinine ≤ 1.5 X upper limit of normal (ULN) OR measured or calculated creatinine clearance (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance [CrCl]) ≥ 60 mL/min for subject with creatinine levels > 1.5 X institutional ULN
* Serum total bilirubin ≤ 1.5 X ULN OR direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) ≤ 2.5 X ULN OR ≤ 5 X ULN for subjects with liver metastases
* Albumin ≥ 2.5 mg/dL
* International normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants.
* Activated partial thromboplastin rime (aPTT) ≤ 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants.
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication; if the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication; subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
* Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Exclusion Criteria:

* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment, patients with human immunodeficiency virus (HIV) adequately controlled on antiretrovirals (undetectable viral load) and patients with chronic lymphocytic leukemia (CLL) not requiring systemic treatment will be included; in addition, steroids for physiologic replacement will be allowed (must be equal to or less than 10mg of prednisone/day).
* Has a known history of active TB (bacillus tuberculosis).
* Hypersensitivity to pembrolizumab or any of its excipients.
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study day 1 or who has not recovered (i.e., ≤ grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study day 1 or who has not recovered (i.e., ≤ grade 1 or at baseline) from adverse events due to a previously administered agent.

  * Note: subjects with ≤ grade 2 neuropathy are an exception to this criterion and may qualify for the study.
  * Note: if subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* Has a known additional malignancy that is progressing or requires active treatment; exceptions include basal cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer. Asymptomatic CLL, not requiring intervention will be included as long as patients meet routine laboratory parameters of the study as outlined above. In addition, patients who have undergone curative bone marrow transplant and currently not requiring immunosuppression, will be allowed on study.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis; subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment; this exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs); replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis.
* Has an active infection requiring systemic therapy; exception HIV on antiretrovirals with negative viral load.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Has received prior therapy with an anti-programmed cell death (PD)-1, anti- programmed cell death 1 ligand (PD-L)1, or anti-PD-L2 agent.
* Has known active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] is detected).
* Has received a live vaccine within 30 days of planned start of study therapy. Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist) are live attenuated vaccines, and are not allowed.
* cSCC that is curable via radiation or surgery; palliative radiation is allowed as long as measurable disease outside radiation field is present for study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-01-27 (Actual); Primary Completion 2021-05-18 (Actual); Study Completion 2021-05-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lowe, MD, MA, Principal Investigator — Emory University
Locations (1):
- Emory University/Winship Cancer Institute, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Pembrolizumab: Patients receive pembrolizumab IV over 30 minutes on day 1. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Pembrolizumab
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: all participants except patient diagnosed with covid
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 11
Age, Continuous [Median (Full Range); unit: years] | 67 [46 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Response Rate of Pembrolizumab
Description: Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: Up to 1 year after treatment discontinuation (max treatment duration of 3 years)
Population: all patients except patient diagnosed with covid-19
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Pembrolizumab)
Number analyzed (Participants) | 11
percentage of participants | 72.73 [39.03 to 93.98]

2. Secondary Outcome: Overall Survival
Description: Number of patients who were alive 1 year after their respective treatment completion dates
Time Frame: Up to 1 year after treatment discontinuation (max treatment duration of 3 years)
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 11
Participants | 11

3. Secondary Outcome: Progression-free Survival
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: Up to 6 months after treatment discontinuation (max treatment duration of 3 years)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 11
percentage of participants | 81.8 [44.7 to 95.1]

ADVERSE EVENTS:
Time Frame: 1 year after treatment discontinuation (max treatment duration of 3 years)
Arm/Group | Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 6/11
Other Adverse Events (participants affected / at risk) | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pembrolizumab (N=11)
Edema cerebral (Nervous system disorders) | 1
Fall (Musculoskeletal and connective tissue disorders) | 1
General disorders and administration site conditions - Other, specify (Injury, poisoning and procedural complications) | 1
Hematoma (Injury, poisoning and procedural complications) | 1
Hydrocephalus (Nervous system disorders) | 1
Hypotension (Cardiac disorders) | 1
Meningitis (Nervous system disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Presyncope (Cardiac disorders) | 1
Seizure (Nervous system disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pembrolizumab (N=11)
Hyperglycemia (Endocrine disorders) | 9
Hyponatremia (Endocrine disorders) | 7
Anemia (Blood and lymphatic system disorders) | 5
Creatinine increased (Hepatobiliary disorders) | 5
Diarrhea (Gastrointestinal disorders) | 4
Activated partial thromboplastin time prolonged (Cardiac disorders) | 4
Aspartate aminotransferase increased (Hepatobiliary disorders) | 4
Blood bilirubin increased (Hepatobiliary disorders) | 4
Fatigue (General disorders) | 4
Alanine aminotransferase increased (Hepatobiliary disorders) | 3
Alkaline phosphatase increased (Hepatobiliary disorders) | 3
Dry mouth (General disorders) | 3
Dyspnea (Gastrointestinal disorders) | 3
Headache (Nervous system disorders) | 3
Hyperkalemia (Cardiac disorders) | 3
Hypertension (Cardiac disorders) | 3
Hyperuricemia (Gastrointestinal disorders) | 3
Hypoalbuminemia (Blood and lymphatic system disorders) | 3
Hypocalcemia (Cardiac disorders) | 3
Hypoglycemia (Endocrine disorders) | 3
Hypomagnesemia (Cardiac disorders) | 3
Pain (General disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 3
Anorexia (Gastrointestinal disorders) | 2
Bruising (Injury, poisoning and procedural complications) | 2
Constipation (Gastrointestinal disorders) | 2
Cough (Infections and infestations) | 2
Dysphagia (Musculoskeletal and connective tissue disorders) | 2
Fall (Musculoskeletal and connective tissue disorders) | 2
Flu like symptoms (Infections and infestations) | 2
General disorders and administration site conditions - Other, specify (General disorders) | 2
Hemoglobin increased (Blood and lymphatic system disorders) | 2
Hypermagnesemia (Cardiac disorders) | 2
Hypokalemia (Blood and lymphatic system disorders) | 2
Hypothyroidism (Endocrine disorders) | 2
Insomnia (Psychiatric disorders) | 2
Metabolism and nutrition disorders - Other, specify (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 2
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 2
Platelet count decreased (Blood and lymphatic system disorders) | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Urine discoloration (Renal and urinary disorders) | 2
Adrenal insufficiency (Hepatobiliary disorders) | 1
Allergic reaction (Immune system disorders) | 1
Aspiration (Injury, poisoning and procedural complications) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1
Blurred vision (Eye disorders) | 1
Chills (General disorders) | 1
Depression (Psychiatric disorders) | 1
Dizziness (General disorders) | 1
Edema cerebral (Nervous system disorders) | 1
Edema limbs (Blood and lymphatic system disorders) | 1
Fever (Infections and infestations) | 1
Flushing (Blood and lymphatic system disorders) | 1
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1
Hematoma (Blood and lymphatic system disorders) | 1
Hydrocephalus (Nervous system disorders) | 1
Hypercalcemia (General disorders) | 1
Hypernatremia (Blood and lymphatic system disorders) | 1
Hypophosphatemia (Congenital, familial and genetic disorders) | 1
Hypotension (Cardiac disorders) | 1
Infections and infestations - Other, specify (Infections and infestations) | 1
Investigations - Other, specify (General disorders) | 1
Laryngeal hemorrhage (Ear and labyrinth disorders) | 1
Laryngeal inflammation (Ear and labyrinth disorders) | 1
Meningitis (Nervous system disorders) | 1
Movements involuntary (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Palpitations (Cardiac disorders) | 1
Papulopustular rash (Skin and subcutaneous tissue disorders) | 1
Paresthesia (Nervous system disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 1
Postnasal drip (Ear and labyrinth disorders) | 1
Presyncope (General disorders) | 1
Seizure (Nervous system disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1
Skin ulceration (Skin and subcutaneous tissue disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Thromboembolic event (Blood and lymphatic system disorders) | 1
Vaginal hemorrhage (Reproductive system and breast disorders) | 1
Vascular disorders - Other, specify (Musculoskeletal and connective tissue disorders) | 1
Ventricular arrhythmia (Blood and lymphatic system disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Weight loss (General disorders) | 1
White blood cell decreased (Blood and lymphatic system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-12-13): https://cdn.clinicaltrials.gov/large-docs/59/NCT02964559/Prot_SAP_001.pdf
  • Informed Consent Form (2019-09-11): https://cdn.clinicaltrials.gov/large-docs/59/NCT02964559/ICF_000.pdf